CLINICAL TRIAL: NCT04466722
Title: A-LIST What Matters Most Insights Series
Brief Title: The A-LIST WMM Insights Series
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UsAgainstAlzheimer's (Other)
Responsible Party: Sponsor
Other Study IDs: A-LIST Protocol 1
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Alzheimer Disease; Dementia; Mild Cognitive Impairment
Keywords: Alzheimer; Dementia; Cognitive; Cognition; Brain health
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of the Study is to develop an understanding over time and through multiple research projects, including surveys, interviews, online focus groups, and other primary research methodologies (A-LIST Research Projects) on what matters most to individuals concerned about brain health and those with and/or affected by Alzheimer's disease and other dementias, including caregivers.

DETAILED DESCRIPTION:
To do this, UsAgainstAlzheimer's will identify and engage individuals who want to focus on brain health; individuals who are worried about their cognition; individuals who perceive themselves to be at risk for Alzheimer's disease (AD); individuals who may be at risk for AD due to self-identified confirmation of underlying disease pathology; individuals who self-identify as having a diagnosis of mild cognitive impairment (MCI) or of AD or another dementia; and those who self-identify as current or former caregivers of patients with Alzheimer's disease or another dementia to participate in the A-LIST Research Projects. Such participants will either already be - or will be invited to become - members of the A-LIST cohort, an online cohort of individuals ready and willing to engage in A-LIST WMM Insights Series (A-LIST members).

The A-LIST WMM Insights Series will enlist participants to offer insights into a range of issues relevant to Alzheimer's, including as examples issues pertinent to clinical trial design, regulatory submissions, other research strategies, payer value determinations, and care and services research. The A-LIST WMM Insights Series may seek information that in some instances will be marketing research or other research exempt from IRB oversight. However, when an individual A-LIST Research Project constitutes human subjects research consistent with governing law, IRB approval will be sought and obtained. Where questions exist whether an individual A-LIST Research Project constitutes human subject research, IRB determination will be solicited.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in the Study, an individual must meet all of the following criteria:

1. Age 18 years or older.
2. United States, Canada resident.
3. Self-report of cognitive difficulties, caregiver status or interest in brain health.
4. Have indicated willingness to participate by selecting "I Agree" option when joining the A-LIST. Additionally, will have clicked on link - invitation to take a specific survey
5. Able to speak, read, and understand English.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this Study:

1. Unable to comply with the Study requirements.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who want to focus on brain health; individuals who are worried about their cognition; individuals who perceive themselves to be at risk for Alzheimer's disease (AD); individuals who may be at risk for due to self-identified confirmation of underlying disease pathology; individuals who self-identify as having a diagnosis of mild cognitive impairment (MCI) or of AD or another dementia; and those who self-identify as current or former caregivers of patients with Alzheimer's disease or another dementia.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Phenotypical Characteristics of Patients and Caregivers | 3 years
  Online monthly surveys capture the burden and unmet needs for patients and caregivers of individuals with or at risk for Alzheimer's disease, other dementias, and mild cognitive impairment; also recruiting individuals interested in brain health.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Frangiosa, MBA, Principal Investigator — UsAgainstAlzheimer's
Locations (1):
- UsAgainstAlzheimer's, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Join UsAgainstAlzheimer's A-LIST — https://www.usagainstalzheimers.org/networks/A-LIST